CLINICAL TRIAL: NCT02486861
Title: OCT-Features Of moRphology, coMposItion anD instABility of Culprit and Not Culprit Coronary pLaquE in ACS Patients
Brief Title: OCT-Features in Culprit and Not Culprit Coronary Plaque in ACS Patients
Acronym: OCT-FORMIDABLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Mario Iannaccone, M.D. Cardiology Fellow, A.O.U. Città della Salute e della Scienza
Other Study IDs: 349/2015
Record Dates: First submitted 2015-06-24; First posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Acute Coronary Syndrome; Culprit Plaque; Non Culprit Plaque
Keywords: Tomography, Optical Coherence
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- culprit plaque: correlation of OCT characteristics of culprit plaque with incidence of major adverse cardiovascular events (MACEs defined as the composite of death from cardiac causes, non- fatal MI, clinically driven target vessel revascularization (TVR), or re-hospitalization due to unstable or progressive angina according to Braunwald Unstable Angina Classification) and clinical baseline characteristics.
  Interventions: Other: optical coherence tomography
- non culprit plaque: correlation of OCT characteristics of non culprit plaque of culprit plaque with incidence of major adverse cardiovascular events (MACEs defined as the composite of death from cardiac causes, non- fatal MI, clinically driven target vessel revascularization (TVR), or re-hospitalization due to unstable or progressive angina according to Braunwald Unstable Angina Classification) and clinical baseline characteristics.
  Interventions: Other: optical coherence tomography

INTERVENTIONS:
Other: optical coherence tomography

SUMMARY:
The OCT-FORMIDABLE register will include with a retrospective fashion all consecutive patients that perform OCT on culprit and not culprit plaque in any subset in patients with ACS. Clinical and OCT data will be included in the register according to the dataset.The primary endpoint will be the correlation of OCT characteristics with incidence of major adverse cardiovascular events (MACEs defined as the composite of death from cardiac causes, non- fatal MI, clinically driven target vessel revascularization (TVR), or re-hospitalization due to unstable or progressive angina according to Braunwald Unstable Angina Classification) and clinical baseline characteristics.

In particular subanalysis will be performed in the following subgroups: culprit plaque, not culprit plaque in culprit vessel, not culprit plaque in different vessel.

Secondary end-point will be to evaluate how OCT analysis changed interventional cardiology approach in culprit plaque definition and coronary stenting respect the coronary angiography alone.

DETAILED DESCRIPTION:
INTRODUCTION. Pathophysiology of Acute Coronary Syndrome (ACS) deeply differs from those of stable patients, mainly due to peculiar features of plaque. Interestingly, most of the lesions triggering an acute ischemic event, usually defined "culprit lesions" are not angiographically severe, but present with mild stenosis. However, when evaluated at autopsy or with intracoronary imaging, they show often a pro-thrombotic pattern, with thin cap fibroatheroma, soft plaques and thrombus, prone to rupture.

Patients without culprit plaque rupture (CPR) exhibit different mechanisms of instability including thrombus at the site of plaque erosion, or intense vasoconstriction of epicardial arteries or coronary microcirculation disfunction.

In this setting, in the last years Optical Coherence Tomography (OCT) has emerged as the most accurate instrument for intracoronary evaluation. Due to a resolution of approximately 10-20 µm it has been largely exploited in the evaluation and characterization of plaque features, both in stable and acute coronary artery disease.

On the other hand, despite recent evidences, characteristics of culprit plaque in different subset of patients are not well defined. Moreover clinical significance of plaque characteristics is unknown.

METHODS The OCT-FORMIDABLE register will include with a retrospective fashion all consecutive patients that perform OCT on culprit and not culprit plaque in any subset in patients with ACS. Clinical and OCT data will be included in the register according to the dataset.

SAMPLE SIZE: the recent paper of Niccoli et al showed a percentages of plaque rupture of 60% in ACS. According to the paper by Pedruzzi et al, at least 100 patients are needed to evaluate independent predictive power of clinical presentation (STEMI vs NSTEMI vs UA), diabetes mellitus, previous use of aspirin, of statin and age.

OCT ANALYSIS Different OCT system analysis and technique (different pullback velocity 75 mm vs 54 mm, contrast mediated or ringer lactate injection) will be reported. Each center will evaluate the OCT image by internal committee composed by at least two people. In case of discordance an external opinion will be required.

Plaque rupture will be defined as the presence of fibrous cap discontinuity leading to a communication between the inner (necrotic) core of the plaque and the lumen. Plaque rupture included also fibrous cap disruption detected over a calcified plaque characterized by protruding calcification, superficial calcium, and the presence of substantive calcium proximal or distal to the lesion.

Thin cap fibro atheroma will be defined as cap thickness < 65 nm. Thin cap fibro atheroma at rupture site will be reported.

Fibrocalcific, fibrotic plaque, lipid component or macrophage infiltration will be defined according to the recent proposed criteria and reported.

Data will be divided according the clinical significance of the studied plaque, in particular culprit plaque, not culprit plaque in culprit vessel and not culprit plaque in other vessels.

Moreover will be recoded if OCT analysis changed the interventional cardiologist approach in deciding the culprit lesion to treat.

CLINICAL FOLLOW-UP AND ENDPOINT DEFINITION A clinical follow-up at least of 12 months after discharge will be evaluated.

The primary endpoint will be the correlation of OCT characteristics with incidence of major adverse cardiovascular events (MACEs defined as the composite of death from cardiac causes, non- fatal MI, clinically driven target vessel revascularization (TVR), or re-hospitalization due to unstable or progressive angina according to Braunwald Unstable Angina Classification) and clinical baseline characteristics.

In particular subanalysis will be performed in the following subgroups: culprit plaque, not culprit plaque in culprit vessel, not culprit plaque in different vessel.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients that perform OCT on culprit and not culprit plaque in any subset in patients with ACS.

Exclusion Criteria:

* low quality OCT images
* cardiogenic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The OCT-FORMIDABLE register will include with a retrospective fashion all consecutive patients that perform OCT on culprit and not culprit plaque in any subset in patients with ACS. Clinical and OCT data will be included in the register according to the dataset.
  SAMPLE SIZE: the recent paper of Niccoli et al11 showed a percentages of plaque rupture of 60% in ACS. According to the paper of Pedruzzi et al12, at least 100 patients are needed to evaluate independent predictive power of clinical presentation (STEMI vs NSTEMI vs UA), diabetes mellitus, previous use of aspirin, of statin and age.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
the correlation of OCT characteristics with incidence of major adverse cardiovascular events (MACEs) and clinical baseline characteristics. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Iannaccone, Turin, Turin, Italy

REFERENCES:
- [Derived] Giordana F, Errigo D, D'Ascenzo F, Montefusco A, Garbo R, Omede P, D'Amico M, Moretti C, Tamburino C, Ferrari GM. Female sex impact on culprit plaque at optical coherence tomography analysis in the setting of acute coronary syndrome in OCT-FORMIDABLE registry. Future Cardiol. 2020 Mar;16(2):123-131. doi: 10.2217/fca-2018-0073. Epub 2020 Jan 22. PMID 31965820
- [Derived] Iannaccone M, Souteyrand G, Niccoli G, Mancone M, Sardella G, Tamburino C, Templin C, Gili S, Boccuzzi GG, D'Ascenzo F. Clinical impact of optical coherence tomography findings on culprit plaque in acute coronary syndrome: The OCT-FORMIDABLE study registry. Catheter Cardiovasc Interv. 2018 Dec 1;92(7):E486-E492. doi: 10.1002/ccd.27633. Epub 2018 May 10. PMID 29745476
- See also: Related Info — http://www.cardiogroup.org